CLINICAL TRIAL: NCT04958044
Title: Endoscopic Assisted Calcium Electroporation in Esophageal Cancer - a Safety Study
Brief Title: Endoscopic Assisted Calcium Electroporation in Esophageal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Patrick Achiam (Other)
Responsible Party: Sponsor-Investigator, Michael Patrick Achiam, Consultant, Ass. Professor, MD, DMSci, Ph.D., FEBS-OG, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: eCaEP2021
Record Dates: First submitted 2021-06-24; First posted 2021-07-12 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Calcium Gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Calcium electroporation (Experimental): Calcium gluconate 0.23 mmol/ml Maxium dosage 20 ml Intra tumoral injection
  Interventions: Drug: Calcium Gluconate

INTERVENTIONS:
Drug: Calcium Gluconate — Calcium electroporation

SUMMARY:
In this pilot study, patients with non-curable esophageal cancer will be treated with endoscopic assisted calcium electroporation (CaEP). CaEP is a novel cancer treatment where intratumoral injection with calcium is combined with locally applied electrical pulses, in order to increase calcium influx which leads to tumor necrosis.

It is hypothesized that:

* Endoscopic assisted CaEP is a safe and feasible procedure in patients with non-curable esophageal cancer
* CaEP debulks the tumor, facilitating the patient's ability to eat and drink

In this single-arm pilot study, eight patients will be treated.

DETAILED DESCRIPTION:
Electroporation facilitates the transport of molecules across the cell membrane and into the cell by means of electrical pulses. An electric field applied to the cell destabilizes the cell membrane forming cracks, which reseals after a few minutes. During this time slot, molecules which normally are impermeable to the cell membrane are able to cross into the cytosol of the cell. Within the last ten years, studies have shown that the combination of intratumoral injection of calcium and electroporation (Calcium electroporation/CaEP) is an effective method in killing cancer cells. CaEP has been evaluated in clinical studies in colorectal cancer, carcinomas in the head and neck area, and in cutaneous metastases with promising results.

In this single-arm pilot study, eight patients with non-curable esophageal cancer will be included.

It is hypothesized that:

* Endoscopic assisted CaEP is a safe and feasible procedure in patients with non-curable esophageal cancer
* CaEP debulks the tumor, facilitating the patient's ability to eat and drink
* CaEP induces a systemic immunological response

The primary objective is to evaluate the safety of CaEP for esophageal cancer. Adverse Events (AE) and Serious Adverse Events (SAE) will be evaluated.

Secondary outcomes include:

* dysphagia (Mellow Pinkas dysphagia score)
* pain (Numeric Rating Scale, NRS)
* quality of life (QoL) (EORTC QLQ-C30)
* tumor response evaluated from computed tomography (CT) and upper endoscopy
* immunologic response

Tertiary outcomes include:

✓ 90-days survival

Participants are initially treated once according to protocol. If well-tolerated, the treatment can be repeated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years old.
2. Histological verified malignant tumor in the esophagus.
3. Subjects must have been considered unsuitable for potential curative treatment.
4. Locally progressive disease, and other standard oncological treatment have been administrated and/or considered first.
5. Performance status ECOG/WHO < 2.
6. Expected survival > 3 months.
7. Platelets ≥ 50 billion/l, International Normalized Ratio (INR) < 1,5.
8. Subjects must be willing and able to comply with the procedure such as agreed follow-up visits.
9. Women of childbearing potential (WOCBP) and male partners to WOCBP should use adequate contraception during the trial.
10. Subjects must give written informed consent.

Exclusion Criteria:

1. Coagulation disorder that cannot be corrected.
2. Subjects with a clinically significant cardiac arrhythmia.
3. Pregnancy or lactation.
4. Concurrent treatment with another investigational medicinal product.
5. Stenosis that prevents passage of the endoscope with the device attached.
6. Patients with any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Safety | 14 days after treatment
  Registration of all AE/SAE´s within the first 14 days after treatment. The events will be assessed by CTCAE v4.0.

SECONDARY OUTCOMES:
Dysphagia | After 7 days, 2-4 weeks and after 6-8 weeks.
  According to Mellow Pinkas dysphgia scale
Pain | After 7 days, 2-4 weeks and after 6-8 weeks.
  Assesed by Numerical Rating Scale
Qualitiy of life | After 7 days, 2-4 weeks and after 6-8 weeks.
  Assesed by "EORTC QLQ-C30"
90 days survival | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Egeland C, Baeksgaard L, Gehl J, Gogenur I, Achiam MP. Palliative Treatment of Esophageal Cancer Using Calcium Electroporation. Cancers (Basel). 2022 Oct 27;14(21):5283. doi: 10.3390/cancers14215283. PMID 36358702